CLINICAL TRIAL: NCT03066284
Title: A Qualitative Study on the Experiences and Expectations of Children and Adolescents Having Type 1 Diabetes Towards Insulin Pump Therapy and Its Effect on Their Quality of Life in Kuwait
Brief Title: A Qualitative Study on CSII in Children and Adolescents Having Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, nehad Taha, Senior Diabetes Educator, Dasman Diabetes Institute
Other Study IDs: RA 2016-006
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Children; Adolescents; Parents; Insulin Pump Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Using qualitative method; a qualitative case study using semi-structured interviews to explore patients' experiences. Study population of insulin pump patients aged 11-18 years old will be recruited from pediatrics with T1D at Dasman Diabetes Institute; who started using CSII at least one year ago and their parents. Semi-structured interviews will be recorded and then transcribed word by word. Data analysis will be performed using an inductive thematic approach.

DETAILED DESCRIPTION:
SPECIFIC AIMS

1. To explore the experiences of adolescents and their parents and parents ofi children with type 1 diabetes in Kuwait about the use of Insulin Pump Therapy (IPT) in the context of their quality of life.
2. To gain in-depth understanding of the perceptions of adolescents and their parents and parents of children with type 1 diabetes in Kuwait with T1DM about IPT and its use for diabetes management.

Design A qualitative case study methodology will be adopted using semi-structured interviews for data gathering. Interviews will be conducted with a purposive sample including adolescents and their parents and parents of children with type 1 diabetes in Kuwait with T1D, who are on CSII therapy at least 12 months, along with their parents.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1 D in Kuwait as specified by their Consultant and in line with the Kuwait Clinical Guidelines diagnosis of T1D (2006) criteria
* Adolescents between the age of 11 and 18 or children between 2 and 10 years old
* Kuwaiti or expats
* Duration of CSII (Insulin Pump Therapy) at least 12 months.
* Prior to starting Insulin Pump Therapy must have been on MDI for a minimum of 12 months
* Attend the Insulin Pump clinic at DDI

Exclusion Criteria:

* Non-English & non-Arabic speakers
* Presence of a learning disability
* Diagnosis of any diabetes complication before starting the CSII therapy
* Diagnosis of psychological problem

Ages: 4 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: adolescents and their parents and parents of children with type 1 diabetes in Kuwait with T1D, who are on CSII therapy at least 12 months, and were on MDI for at least 12 months before initiation of CSII
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-03-14 (Actual); Primary Completion 2017-03-13 (Estimated); Study Completion 2019-03-13 (Estimated)

PRIMARY OUTCOMES:
Impact of IPT on QoL of children and adolescents from their perspective and their parents' perspective | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A. Taha, MSc., Principal Investigator — Dasman Diabetes Institute; Naglaa I. Mesbah, MSc., Principal Investigator — Dasman Diabetes Institute; Zahra N. Rahme, MSc., Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Sharq, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No